CLINICAL TRIAL: NCT01385917
Title: Study of Clinical and Radiological Changes in Patients With Duchenne Muscular Dystrophy Theoretically Treatable With Exon 53 Skipping
Brief Title: Observational Study of Patients With Duchenne Muscular Dystrophy Theoretically Treatable With Exon 53 Skipping
Acronym: pre U7-53
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Genethon (Other)
Collaborators: Institute of Myology (Other)
Responsible Party: Sponsor
Other Study IDs: GHN007.10
Record Dates: First submitted 2011-06-29; First posted 2011-06-30 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-03

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; strength and function tests; MRI
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Total blood count with differential leukocyte count Assay of immunoglobulins and the various sub-classes (IgG, IgM, IgA, IgE) Test for immunisation against all AAV serotypes Serum urea, creatinine, AST/ALT , GammaGT, bilirubin, CK, alkalin phosphatase
Oversight: Data Monitoring Committee: No

SUMMARY:
PreU7-53 is a natural history study. The objective is to monitor the clinical and radiological course of upper limb muscle impairment in patients with Duchenne Muscular Dystrophy (DMD), potentially treatable with AAV-mediated exon 53 skipping.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Duchenne muscular dystrophy confirmed by at least genetic testing, theoretically treatable by exon 53 skipping.
* Age between ≥ 12 and <20 years old.
* Non ambulant patients (i;e; inability to walk more than 10 meters without any of assistance).
* Patients covered by a national health insurance scheme.
* Signed informed consent.

Exclusion Criteria:

* Patient incapable of sitting upright in a wheelchair for at least one hour.
* Patients with severe intellectual impairment preventing them from fully understanding the exercises to be performed.
* Recent (less than 6 months ago) upper limb surgery or trauma This criteria is however no definitive. Patients who have undergone upper limb surgery or trauma may nonetheless be enrolled once the 6 month period is over.
* Known immune deficiency.
* Contraindications to NMR exams

Ages: 12 Years to 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with theoretically exon 53 skipping-treatable DMD
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2011-10; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
PreU7-53 is a natural history study | Every year
  The objective is to monitor the clinical and radiological course of upper limb muscle impairment in patients with DMD, potentially treatable with AAV-mediated exon 53 skipping.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent SERVAIS, MD, Principal Investigator — Myology Institute
Locations (2):
- Myology Institute, Paris, France
- Great ormond Street Hospital & University College London Hospital, London, United Kingdom